CLINICAL TRIAL: NCT03588650
Title: A Phase 1 Study of HLX20, a Human Monoclonal Antibody Targeting Programmed Death Ligand 1 (PD-L1) Protein in Patients With Advanced Solid Tumors
Brief Title: A Phase 1 Study of HLX20, a Human Monoclonal Antibody Targeting PD-L1Protein in Patients With Advanced Solid Tumors
Acronym: HLX20
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HLX20-001
Record Dates: First submitted 2018-06-22; First posted 2018-07-17 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX20, in patients with solid tumors (Experimental): Each cycle of treatment consists of 4 weeks. Patients who enroll into this study will receive an infusion of assigned dose of HLX20 once every two weeks. No intra-patient dose escalation is allowed. The proposed dose escalation sequence is 1, 3, 10 and 20 mg/kg, starting from 1 mg/kg.
  Interventions: Drug: HLX20

INTERVENTIONS:
Drug: HLX20 — a Human Monoclonal Antibody Targeting Programmed Death Ligand-1 (PD-L1) Protein

SUMMARY:
This is an open-label, dose escalation, first-in-human study of HLX20, an anti-PD-L1 monoclonal antibody, in patients with metastatic or recurrent solid tumors who have failed standard therapy.

DETAILED DESCRIPTION:
Tumor microenvironment plays an important role in the interaction of immune cells with cancer . The identification of programmed cell death receptor 1 (PD-1) and programmed death ligand-1 (PD-L1) have provided the scientific rationale and supports the clinical development of agents targeting this pathway. Currently, PD-1 and PD-L1 inhibitory pathway blockade has demonstrated impressive activity against a spectrum of multiple tumor types, including Hodgkin's lymphoma, melanoma, bladder cancer, lung cancer, renal cell carcinoma.

HLX20 is a novel anti-PD-L1 monoclonal antibody. In the nonclinical pharmacology studies, HLX20 has demonstrated anti-tumor activities in xenogenic animal models comparable to currently available anti-PD-L1 monoclonal antibodies. HLX20 binds to PD-1 and PD-L1 inhibitory pathway and human PD-L1 at high affinity, and mouse PD-L1 at much lower affinity. HLX20 does not cause hemolysis to human red blood cells and has no local irritation to human tissues. (The results of pharmacokinetic (PK)/toxicokinetic studies in cynomolgus studies have been described in detail in the Investigator's Brochure.)The no-observable adverse effect level (NOAEL) is set at 100 mg/kg every 2 weeks for 13 weeks in cynomolgus studies.

Based on these results, the initial dose 1 mg/kg every 2 weeks was chosen for this study .This dose level is approximately 30-fold lower than the human equivalent dose of NOAEL from preclinical toxicology studies. An adaptive Bayesian dose-finding design will be used to identify the MTD (maximum tolerated dose). The target toxicity rate for the MTD is set at 0.3 and the maximum sample size is 30.The safety profiles at different dose levels, PK parameters, biomarkers, pharmacodynamic markers, immunogenicity as well as the preliminary efficacy of the drug, will also be investigated in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females of 18 years of age or older (or per local regulations).
2. Have histologically-proven measurable, or evaluable advanced (systemically or locally progressive), or metastatic solid tumors or the locally advanced disease is not amenable to local therapy, who have failed, or are intolerant to standard therapy or for whom no standard therapy is available. (For patients with hepatocellular carcinoma, the diagnosis needs to be supported by dynamic computed tomography [CT]/magnetic resonance imaging, if pathological confirmation is not attainable).
3. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2 at the time of study entry.
4. Able to comprehend and provide informed consent.
5. A life expectancy longer than 3 months in the opinion of the Investigator.
6. Adequate hematologic functions, as defined by: absolute neutrophil counts

   ≥ 1500/mm3; a hemoglobin level ≥ 10 g/dL; a platelet count ≥ 100,000/mm3.
7. Adequate hepatic function defined by: a total bilirubin level ≤ 1.5 × of upper limit of normal (ULN); aspartate transaminase and alanine transaminase levels ≤ 2.5 × ULN or ≤ 5 × ULN in known hepatic metastases or with primary hepatocellular carcinoma.
8. Adequate renal function, as defined by the creatinine clearance ≥ 50 mL/minute (as calculated by the Cockcroft-Gault formula).
9. Adequate cardiac function defined as left ventricular ejection fraction ≥ 50% by cardiac ultrasound or multigated acquisition (MUGA) scan. A recent MUGA scan is acceptable if performed within 8 weeks of the first infusion of IP.
10. Females of child-bearing potential must have a negative pregnancy test upon entry into this study and must be willing to use highly effective birth control upon enrollment, during the Treatment Phase and for 180 days following the last dose of study drug. A female is considered of child-bearing potential following menarche and until becoming postmenopausal (no menstrual period for a minimum of 12 months) unless permanently sterile (undergone a hysterectomy, bilateral salpingectomy, or bilateral oophorectomy).
11. If male, must be surgically sterile or willing to use highly effective birth control upon enrollment, during the Treatment Phase, and for 180 days following the last dose of study drug.
12. History of prior major surgery, prior cytotoxic chemotherapy, or prior therapy with investigational agents, medical device, or local radiotherapy should be at least 28 days prior to Screening and at least 42 days from the last infusion of immune check point inhibitors (including anti-programmed cell death receptor-1 [PD-1] or anti-PD-L1) before the first infusion of IP.
13. Child-Pugh score of A (patients with hepatocellular carcinoma only).
14. Able to be followed up as required by the study protocol.

Exclusion Criteria:

1. Persistent ≥ Grade 2 toxicities from prior therapies, with the exception of alopecia of any grade, Grade ≤ 2 peripheral neuropathy, and laboratory values listed per the inclusion criteria.
2. Concurrent unstable or uncontrolled medical conditions, including:

   * Active systemic infections;
   * Poorly controlled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg), or poor compliance with antihypertensive agents;
   * Clinically significant arrhythmia, unstable angina pectoris, congestive heart failure (Class III or IV of New York Heart Association) or acute myocardial infarction within 6 months;
   * Uncontrolled diabetes or poor compliance with hypoglycemic agents;
   * The presence of chronically unhealed wound or ulcers;
   * Other chronic diseases, which, in the opinion of the Investigator, could compromise safety of the patient or the integrity of the study.
3. Newly-diagnosed or symptomatic brain metastases (patients with a history of brain metastases must have received definitive surgery or radiotherapy, be clinically stable, and not be taking steroids for brain edema). Anticonvulsants are allowed. Patients with history of leptomeningeal disease will be excluded.
4. Any concurrent malignancy other than basal cell carcinoma or carcinoma in situ of the cervix. (Patients with a previous malignancy but without evidence of disease for ≥ 3 years are allowed to participate).
5. Females who are pregnant, lactating, or intend to become pregnant during their participation in this study.
6. Known history of human immunodeficiency virus infection.
7. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease, diverticulitis with the exception of diverticulosis, celiac disease, irritable bowel disease, Wegner syndrome) within the past 2 years. Patients with well controlled vitiligo, alopecia, and Grave's disease, hypothyroidism (eg, following Hashimoto syndrome) stable on hormone replacement, or psoriasis not requiring systemic treatment (within the past 3 years), or patients with controlled Type 1 diabetes mellitus who are on a stable insulin regimen are not excluded.
8. Current or prior use of immunosuppressive medication within 14 days before the first dose. The following are exceptions to this criterion:

   * Intranasal, inhaled, topical steroids or local steroid injections (eg, intra-articular injection), OR
   * systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, OR
   * steroids as premedication for hypersensitivity reactions (eg, CT scan premedication).
9. History of primary immunodeficiency or allogeneic transplantation.
10. Active hepatitis B (HBsAg reactive). Active hepatitis C virus (HCV) infection, defined as having a positive HCV antibody test followed by a positive HCV RNA test at Screening.
11. History of interstitial lung disease.
12. Receipt of live attenuated vaccines within 30 days prior to the first dose of IP. Patients, if enrolled, should not receive live or live attenuated vaccines during the study and for 30 days after the last dose of IP.
13. The patient is the Investigator, sub-investigator or anyone directly involved in the conduct of the study.
14. History or current evidence of any condition or disease that could confound the results of the study or, in the opinion of Investigator, is not in the best interest of the patient to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-08-07 (Actual); Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of HLX20 in solid tumors patients | 1 year
  The target toxicity rate in this study for the MTD is set at 0.3 ( 30% DLT) identified by an adaptive Bayesian dose-finding design .

SECONDARY OUTCOMES:
Maximum serum concentration (Cmax) of HLX20. | 1 year
Minimum serum concentration (Cmin) of HLX20. | 1 year
Area under serum concentration-time curve within one dosing interval (AUC0-tau) of HLX20. | 1 year
Terminal elimination half-life (T1/2) of HLX20 in different cohorts | 1 year
Clearance rate (CL) of HLX20 | 1 year
Volume of distribution at steady state (Vss) of HLX20. | 1 year
Immunogenicity | 1 year
  The presence and percentage of anti-HLX20 antibody
Disease control rate (DCR) | 1 year
  Number of patients with complete response/partial response/stable disease divided by the total number of patients treated
Overall response rate (ORR). | 1 year
  Number of patients with confirmed complete or partial response, divided by the total number of treated patients with measurable disease at baseline
Receptor occupancy of PD-L1 on human T-cells. | 1 year

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (6):
  - Kinghorn cancer centre, Darlinghurst, New South Wales
  - Macquarie University, Darlinghurst, New South Wales
  - Sunshine Coast University Hospital, Brisbane, Queensland
  - Gold Coast Hospital, Southport, Queensland
  - CMAX Clinical research, Adelaide, South Australia
  - Cabrini Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Undecided